CLINICAL TRIAL: NCT01005017
Title: Percutaneous Radiofrequent Lesioning of the Splanchnic Nerves in Patients With Chronic Pancreatitis
Brief Title: Percutaneous Lesioning Splanchnic Nerves in Patients With Chronic Pancreatitis
Acronym: PRFLSN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Dr. YCA Keulemans, Department of Gastroenterology Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0911111
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Pancreatitis; Chronic Pain; Abdominal Pain
Keywords: Radiofrequent ablation; Percutaneous radiofrequent therapy
MeSH Terms: conditions — Pancreatitis, Chronic; Chronic Pain; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutanous RF lesioning (Active Comparator): Radiofrequent lesioning uses a high frequency alternating current to heat tissues leading to thermal coagulation. It produces predictable and accurate lesions of the splanchnic nerves.
  Interventions: Procedure: Percutaneous Radiofrequent Lesioning
- Optimal medical treatment (No Intervention)

INTERVENTIONS:
Procedure: Percutaneous Radiofrequent Lesioning — One group receives PRFLSN after a positive trial block with bupivacaine, the other group receives no extra treatment besides optimal medical treatment.
  Arms: Percutanous RF lesioning

SUMMARY:
Chronic pancreatitis is a progressive inflammatory disease resulting in slow destruction of the pancreas. This chronic inflammation can lead to chronic abdominal pain which can last for many years. Unfortunately, medical management often is of only limited benefit in treating the pain of chronic pancreatitis.

Management of patients with intractable pain is difficult, often resulting in narcotic addiction.

Early results in a small group of patients suggest that percutaneous radiofrequent lesioning of splanchnic nerves has good potential for pain control in a subset of patients with chronic pancreatitis. Given the simplicity of the procedure, it clearly warrants reappraisal to identify its current role in pancreatic pain management.

DETAILED DESCRIPTION:
Rationale: Pain control is the most pressing problem in patients with chronic pancreatitis. Many methods have been advocated to control this pain. Unfortunately, these methods fail to control the pain in 20-50% of patients. Management of patients with intractable pain is difficult, often resulting in narcotic addiction. Percutaneous alcoholic block of the celiac plexus is, because of the risks of paralysis and catastrophic haemorrhage resulting from injury to major abdominal vasculature, restricted to patients with intractable, severe pain due to terminal pancreatic cancer. Splanchnic nerve lesioning is a useful alternative to celiac plexus block in the management of patients with chronic upper abdominal pain. The predictable relationship of the splanchnic nerves to other structures allows for accurate needle placement and hence a low risk of damage. Radiofrequent lesioning uses a high frequency alternating current to heat tissues leading to thermal coagulation. It produces predictable and accurate lesions.

Objective: To evaluate the feasibility and efficacy of percutaneous radiofrequent lesioning of splanchnic nerves (PRFLSN) in patients with pain caused by chronic pancreatitis. The primary goal is to determine if a 50% reduction in pain can be achieved for at least 3 months. Secondary objectives are reduction of medication use and improvement of quality of life.

Design: Single blind, prerandomized intervention study. Study population: Patients with pain (NRS>5) caused by chronic pancreatitis, despite optimal medical treatment.

Intervention: One group receives PRFLSN after a positive trial block with bupivacaine, the other group receives no extra treatment besides optimal medical treatment.

Main study endpoints: The percentage of reduction of pain after PRFLSN for a period of at least 3 months and preferably one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pancreatitis presenting with significant abdominal pain of pancreatic origin. Pain will be considered significant if there is at least 1 episode of pain every month requiring analgesics during the preceding 3 months, or at least 1 episode of severe pain requiring hospitalization in the preceding 3 months. Pancreatic pain (NRS-score >5 out of 10), resistant to medical therapy, with a duration of at least three months.

Exclusion Criteria:

* Patients with pseudocysts, bile duct obstruction, duodenal obstruction or pancreatic cancer.
* Age younger than 18 years.
* A noncooperative patient.
* Coagulopathy.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Level of pain reduction after PRFLSN compared to optimal medical treatment alone as determined by numeric rating scales (NRS) | 3 months

SECONDARY OUTCOMES:
Level of pain reduction after PRFLSN compared to optimal medical treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yolande CA Keulemans, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MaastrichUMC, Maastricht, Limburg, Netherlands